CLINICAL TRIAL: NCT01406275
Title: Special Drug Use Investigation for CLAVAMOX® (Amoxicillin/Clavulanate) Pediatrics Dry Syrup (Every Indication Excluded Otitis Media)
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 112283
Record Dates: First submitted 2011-07-26; First posted 2011-08-01 (Estimated); Last update posted 2017-05-16 (Actual); Status verified 2017-05

CONDITIONS: Otitis Maedia
MeSH Terms: interventions — Amoxicillin; Clavulanic Acid

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Pediatrics patients prescribed amoxicillin and clavulanate: Pediatrics patients prescribed amoxicillin and clavulanate for treatment of diseases other than otitis media during study period
  Interventions: Drug: Amoxicillin and clavulanate

INTERVENTIONS:
Drug: Amoxicillin and clavulanate

SUMMARY:
This post-marketing surveillance study of CLAVAMOX® was designed to collect and assess the information on proper use, such as safety and efficacy, under actual use conditions, targeting pediatric Japanese patients with diseases (superficial skin infection, deep skin infection, lymphangitis, lymphadenitis, chronic pyoderma, pharyngitis, laryngitis, tonsillitis, acute bronchitis, cystitis, pyelonephritis) other than otitis media.

("CLAVAMOX" is a trademark of the GlaxoSmithKline group of companies.)

ELIGIBILITY:
Inclusion Criteria:

* Pediatric subjects with diseases of superficial skin infection, deep skin infection, lymphangitis, lymphadenitis, chronic pyoderma, pharyngitis, laryngitis, tonsillitis, acute bronchitis, cystitis and pyelonephritis

Exclusion Criteria:

* Not applicable

Max Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Japanese pediatric patients who have superficial skin infection, deep skin infection, lymphangitis, lymphadenitis, chronic pyoderma, pharyngitis, laryngitis, tonsillitis, acute bronchitis, cystitis, pyelonephritis other than otitis media, and treated with amoxicillin and clavulanate
Sampling Method: Probability Sample
Enrollment: 363 (Actual)
Dates: Start 2008-01; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
The number of incidence of adverse events in Japanese pediatric patients, with diseases other than otitis media, treated with amoxicillin and clavulanate based on prescribing information | 2 months
Clinical symptoms after treatment with amoxicillin and clavulanate | 2 months

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline